CLINICAL TRIAL: NCT03724539
Title: Optimizing PharmacoTherapy In the Multimorbid Elderly in Primary CAre: a Cluster Randomized Controlled Trial (the OPTICA Trial)
Brief Title: Optimizing PharmacoTherapy In the Multimorbid Elderly in Primary CAre: the OPTICA Trial
Acronym: OPTICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Utrecht University (Other); University of Basel (Other); University of Zurich (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: U1111-1181-9400
Record Dates: First submitted 2018-10-17; First posted 2018-10-30 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Multimorbidity; Polypharmacy
Keywords: Drug utilization review; Old age

STUDY DESIGN:
Intervention Model Description: Clusters will be randomized 1:1, to either the intervention arm receiving STRIPA or to the control arm undergoing a sham intervention. Each cluster is defined by one GP.
  The patients assigned to a cluster (i.e. GP) which was allocated to the intervention arm will undergo a systematic pharmacotherapy optimization by their GP using the STRIP assistant and shared decision making. Patients assigned to a cluster that was assigned to the control arm will receive a sham intervention, which consists of a usual medication review by the GP in accordance with usual care and shared decision making.
  This RCT randomizes GPs instead of patients to prevent contamination, which would occur if the same GPs treated patients in the intervention and the control arm simultaneously.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The OPTICA study is partially blinded, with blinding being implemented as follows:
  * Due to the nature of the study intervention participating GPs (care providers) cannot be blinded.
  * Patients remain blinded. They will not be informed to which treatment arm their GP is allocated to, in order to minimize performance and other reporting biases. Despite this, they receive a "high-level description" of the study question and the study procedures.
  * Data collection for primary and secondary outcome analyses will be conducted by blinded study team members.
  * Outcome adjudication (MAI and AOU assessment) will be performed by blinded study team members.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STRIPA intervention (Experimental): GPs in the intervention group will perform a STRIPA analysis for each of their 8-10 patients after the recruitment of the patient into the OPTICA trial, so that the results can be discussed in the next consultation and a shared decision-making can be performed.
  STRIPA is a structured method to perform pharmacotherapy optimization. The STRIPA intervention in the OPTICA trial consists of 4 steps:
  1. recording medication and diagnoses in STRIPA (upload from data from the 'Family medicine ICPC Research using Electronic medical records' (FIRE) database)
  2. structured drug review through the GP based on the STRIPA with the integrated STOPP/START criteria
  3. shared decision-making between GP and patient with possible adaptation of the recommendation
  4. follow-up through study team
  Interventions: Device: STRIPA intervention
- Sham intervention (Sham Comparator): Patients in the control group will receive a sham intervention, which consists of a usual medication review by their GP as well as a shared decision making of the latter.
  Interventions: Other: Sham intervention

INTERVENTIONS:
Device: STRIPA intervention — STRIPA is a Dutch software-based tool for the support of the pharmaceutical analysis by 1) taking into account the predictable adverse medication effects, 2) advising safe and appropriate therapy using established STOPP/START criteria, 3) interaction monitoring, and 4) appropriate dosing in accordance with renal function. It represents a highly efficient and user-friendly software engine, which is capable of individually screening the clinical status and pharmacological therapy of older patients with multimorbidity, which can define optimal drug therapy, and which can highlight the adverse drug reaction risk. A summary of these outputs will be used as STRIPA recommendations, which will, if applicable, be implemented by GPs and patients.
  Prior to the STRIPA medication review, the necessary patient information will be loaded from the FIRE database that contains data from more than 300 Swiss GP practices.
  Arms: STRIPA intervention
Other: Sham intervention — Patients being assigned to the control arm will be treated in accordance with standard care. They will receive a sham intervention, which consists of a usual medication review by their GP and a shared decision making between patient and GP.
  Arms: Sham intervention

SUMMARY:
The objective of this randomized controlled trial (RCT) is to evaluate whether the Systematic Tool to Reduce Inappropriate Prescribing (STRIP), put into practice through the STRIP Assistant (STRIPA) and implemented by general practitioners (GPs), will lead to an improvement in clinical and economic outcomes in patients aged 65 or older with multimorbidity and polypharmacy.

DETAILED DESCRIPTION:
Background:

Policy makers face many challenges, when they plan health care systems to meet the needs of the fast growing elderly population. More than 60% of the elderly suffer from multiple chronic conditions (multimorbidity - commonly defined as ≥3 chronic diseases) and get multiple drugs (polypharmacy - commonly defined as ≥5 regular medications). Multimorbid patients are often excluded from randomized controlled trials (RCT) and consequently most prescribing guidelines address diseases in isolation. Consequently, there is inappropriate prescribing, which results in diminished health states and lower quality of life of the patients.

Older patients usually rely on their general practitioners (GPs) to manage their medications. However, GPs often have limited time to adapt polypharmacy. Reviewing medications and understanding their interactions based on a list of diagnoses and drugs is complex and time consuming. Furthermore, due to the increase of patients with multimorbidity and polypharmacy, medication review especially in patients with many drugs is often neglected. Pilot data from the Netherlands showed that a software-assisted method, called STRIPA, was effective for optimizing pharmacotherapy in primary care. Through the OPTICA trial this tool will now be tested in the Swiss primary care context.

Study design:

The OPTICA trial is a single-site cluster randomized controlled trial (RCT), which will be conducted at the Institute for Primary Health Care of the University of Bern (BIHAM). All study-related tasks will be performed centrally at the BIHAM except for patient recruitment and use of the STRIPA, as these two tasks will be performed in participating GP offices.

The GPs in the intervention group use the STRIP assistant, whereas the GPs in the control group conduct a sham intervention: usual medication review and shared-decision making with patient. STRIPA is designed to optimize drug therapy and to advise on safe and appropriate therapy using STOPP/START criteria (STOPP = 'screening tool of older people's prescriptions'; START = 'screening tool to alert to right treatment'). Patients will be followed for 1 year with follow-up phone calls after 6 and 12 months.

Study objectives:

The primary objective of this study is to assess the effect of pharmacotherapy optimization through STRIPA on the medication appropriateness, which is measured by the medication appropriateness index (MAI) for drug overuse and by the assessment of underutilization (AOU) for drug underuse.

The secondary objective of the OPTICA study is to assess the impact of pharmacotherapy optimization by STRIPA on the parameters listed below (1- 4) as well as to examine the use of the STRIP assistant by GPs (5) and to examine patients' willingness to deprescribe (6):

1. Degree of polypharmacy
2. Degree of over- and underprescribing
3. Number of falls and fractures
4. Quality of life, including pain/discomfort
5. Health economic parameters, including direct costs of the intervention and incremental cost-effectiveness
6. Enablers and barriers faced by GPs when using the STRIP assistant
7. Patients' willingness to deprescribe

Statistical considerations:

40 clusters with a cluster size of 8-10 patients will be included. The primary analysis will be an intention-to-treat (ITT) analysis, whereby all randomised patients will be included in the group they were allocated to.

There will be two co-primary outcomes, the improvement in the MAI score at 12 months, defined as decrease of the score of at least one point, and improvement in the AOU index at 12 months, defined as a reduction of at least one prescribing omission. Both outcomes will be tested separately and success claimed if either test is significant. Adjustment for multiple testing will be performed.

In the primary analysis, the investigators will assess outcomes at the patient level, accounting for the correlated nature of data among GPs by using multilevel mixed-effects models. For the co-primary outcomes, the investigators will present and compare the proportion of patients with improvement of the MAI score and AOU index in the control and intervention groups. The relative difference between groups will be assessed using a mixed-effects logistic model with a random intercept at the GP level in order to account for clustering.

Secondary binary outcomes will be evaluated like the primary outcomes. Secondary continuous outcomes will be analyzed using random-effects linear regression with a random intercept at the GP level. Models will additionally be adjusted for the baseline value as a covariate. Secondary count outcomes will be analyzed using random-effects Poisson regression with a random intercept at the GP level.

Health economic analyses will comprise the assessment i) of resource use and cost differences between the trial arms, ii) the assessment of differences in quality-adjusted lifetime between the trial arms (expressed as quality-adjusted life years [QALYs]), and iii) the assessment of the cost-effectiveness of the intervention in comparison with the comparator, i.e. medication review in accordance with standard care.

ELIGIBILITY:
Inclusion Criteria

* Being a regular patient of participating GP
* Age: 65 years of age or older
* Multimorbidity: 3 or more coexistent chronic conditions defined by 3 distinct International Classification in Primary Care -2 (ICPC-2) codes defined as chronic (O'Halloran et al., 2004) with an estimated duration of 6 months or more, or based on a clinical decision supported by Pharmacost Groups (PCG) for chronic conditions in an algorithm from FIRE
* Polypharmacy: Use of five or more different regular drugs (defined as authorized medications with registration numbers) for more than 30 days before signing the informed consent form

Exclusion Criteria

* Inability to provide informed consent from a patient or to obtain informed consent from a proxy for patients with cognitive impairment
* If the patient is already participating in the a different interventional study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 323 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Patients' medication appropriateness, as measured by two complementary co-primary outcomes: Co-primary outcome #1: change in the Medication Appropriateness Index (MAI) | 12 months
  Medication Appropriateness Index (MAI), assessed at baseline as well as at the 6 and 12 months follow-ups for each chronic medication of the patient. The 10 item version of the MAI will be used, but the cost-effectiveness item will be excluded. The MAI score for each medication will range from 0 to 17.
Patients' medication appropriateness, as measured by two complementary co-primary outcomes: Co-primary outcome #2: change in the Assessment of Underutilization (AOU) | 12 months
  Assessment of Underutilization (AOU), assessed for each of the patients' chronic conditions at baseline as well as at the 6 and 12 months follow-ups. For each chronic condition of the patient, the assessors decided whether there is i) no omission, ii) marginal omission, or iii) omission of indicated medication.

SECONDARY OUTCOMES:
Patients' degree of polypharmacy | 12 months
  Numbers of regular long-term medications taken by patients, assessed at baseline as well as the 6 and 12 months follow-ups.
Patients' degree of overprescribing, as measured by the Medication Appropriateness Index (MAI) | 12 months
  The degree of overprescribing be assessed at baseline as well as at the 6 and 12 months follow-ups. The 10 item version of the MAI will be used. The MAI score for each medication will range from 0 to 18.
Patients' degree of underprescribing, as measured by the Assessment of Underutilization | 12 months
  The degree of underprescribing will be assessed at baseline as well as at the 6 and 12 months follow-ups. For each chronic condition of the patient, the assessors decided whether there is i) no omission, ii) marginal omission, or iii) omission of indicated medication.
Patients' falls and fractures | 12 months
  Number of falls and fractures reported by the patients. Assessed at baseline as well as at the 6 and 12 months follow-ups.
Patients' quality of life measured by 5-level version of the European Quality of Life-5 Dimensions questionnaire (EQ-5D), including pain/discomfort. | 12 months
  Assessed by the 5-level version of the European Quality of Life - 5 Dimensions questionnaire (EQ-5D). Assessed at baseline as well as at the 6 and 12 months follow-ups. The questionnaire consists of 5 questions with 5 possible responses each and a visual analogue scale (0-100). The EQ-5D-5L index resulting from this questionnaire ranges from 0 to 1.
Amount of formal care received by patients | 12 months
  Assessed by looking at number of planned and unplanned care sessions received by a patient. Assessed at baseline as well as at the 6 and 12 months follow-ups.
Amount of informal care received by patients | 12 months
  Assessed by looking at unpaid care by e.g. family members, relatives, friends. Assessed at baseline as well as at the 6 and 12 months follow-ups.
Survival | 12 months
  As measured by number of survivors
Patients' Quality-adjusted life years (QALYs) | 12 months
  Assessment will be done at the end of the trial, when all data was collected.
Patients' medical costs | 12 months
  Direct medical costs during one year. Assessment will be done at the end of the trial, when all data was collected.
Cost-effectiveness of the STRIPA intervention | 12 months
  The cost-effectiveness analysis will be performed by combining clinical data, quality of life data as well as data about the amount of formal and informal care collected within the trial, and unit costs that will stem from external sources.
Percentage of recommendations accepted by general practitioners (GPs) | 12 months
  Quantification of the amount of recommendations generated by the STRIP assistant that have been accepted by GPs. Assessed after all the GPs in the intervention group have used the STRIPA.
Percentage of recommendations rejected by general practitioners (GPs) | 12 months
  Quantification of the amount of recommendations generated by the STRIP assistant that have been rejected by GPs. Assessed after all the GPs in the intervention group have used the STRIPA.
Patient's willingness to deprescribe | Baseline
  The willingness of patients' to deprescribe will be assessed by the "revised Patients' Attitudes Towards Deprescribing" (rPATD) questionnaire. Assessed at baseline. The score will range from 0 to 22 for the patient questionnaire and between 0 and 19 for the caregiver questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Streit, Prof., MD, PhD, Principal Investigator — University of Bern
Locations (1):
- Berner Institut für Hausarztmedizin, BIHAM, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited in the Bern Open Repository and Information System (BORIS) (www.boris.unibe.ch). BORIS allows searching and is indexed by search engines.
  All items are stored with a unique Digital Object Identifier (DOI) that can be referenced in respective publication.
  The whole study database in csv format will be available and it will include readme files, metadata, information about the performed processing and analytical steps, variable definitions, and references to vocabularies used to help secondary users to understand and reuse the data.
  Data will only be shared upon request to the sponsor-investigator. The data is owned by the sponsor-investigators. In case of data sharing, a data sharing agreement between the external party and the sponsor-investigator will need to be agreed on and signed.

REFERENCES:
- [Background] Barry PJ, Gallagher P, Ryan C, O'mahony D. START (screening tool to alert doctors to the right treatment)--an evidence-based screening tool to detect prescribing omissions in elderly patients. Age Ageing. 2007 Nov;36(6):632-8. doi: 10.1093/ageing/afm118. Epub 2007 Sep 19. PMID 17881418
- [Background] Chmiel C, Bhend H, Senn O, Zoller M, Rosemann T; FIRE study-group. The FIRE project: a milestone for research in primary care in Switzerland. Swiss Med Wkly. 2011 Jan 28;140:w13142. doi: 10.4414/smw.2011.13142. eCollection 2011. PMID 21279858
- [Background] Gallagher P, O'Mahony D. STOPP (Screening Tool of Older Persons' potentially inappropriate Prescriptions): application to acutely ill elderly patients and comparison with Beers' criteria. Age Ageing. 2008 Nov;37(6):673-9. doi: 10.1093/ageing/afn197. Epub 2008 Oct 1. PMID 18829684
- [Background] Gallagher PF, O'Connor MN, O'Mahony D. Prevention of potentially inappropriate prescribing for elderly patients: a randomized controlled trial using STOPP/START criteria. Clin Pharmacol Ther. 2011 Jun;89(6):845-54. doi: 10.1038/clpt.2011.44. Epub 2011 Apr 20. PMID 21508941
- [Background] Jadad AR, To MJ, Emara M, Jones J. Consideration of multiple chronic diseases in randomized controlled trials. JAMA. 2011 Dec 28;306(24):2670-2. doi: 10.1001/jama.2011.1886. No abstract available. PMID 22203536
- [Background] Meulendijk M, Spruit M, Drenth-van Maanen C, Numans M, Brinkkemper S, Jansen P. General practitioners' attitudes towards decision-supported prescribing: an analysis of the Dutch primary care sector. Health Informatics J. 2013 Dec;19(4):247-63. doi: 10.1177/1460458212472333. PMID 24255051
- [Background] Meulendijk MC, Spruit MR, Willeboordse F, Numans ME, Brinkkemper S, Knol W, Jansen PA, Askari M. Efficiency of Clinical Decision Support Systems Improves with Experience. J Med Syst. 2016 Apr;40(4):76. doi: 10.1007/s10916-015-0423-z. Epub 2016 Jan 20. PMID 26791992
- [Background] Samsa GP, Hanlon JT, Schmader KE, Weinberger M, Clipp EC, Uttech KM, Lewis IK, Landsman PB, Cohen HJ. A summated score for the medication appropriateness index: development and assessment of clinimetric properties including content validity. J Clin Epidemiol. 1994 Aug;47(8):891-6. doi: 10.1016/0895-4356(94)90192-9. PMID 7730892
- [Background] Somers A, Mallet L, van der Cammen T, Robays H, Petrovic M. Applicability of an adapted medication appropriateness index for detection of drug-related problems in geriatric inpatients. Am J Geriatr Pharmacother. 2012 Apr;10(2):101-9. doi: 10.1016/j.amjopharm.2012.01.003. Epub 2012 Feb 1. PMID 22304791
- [Background] O'Mahony D, O'Sullivan D, Byrne S, O'Connor MN, Ryan C, Gallagher P. STOPP/START criteria for potentially inappropriate prescribing in older people: version 2. Age Ageing. 2015 Mar;44(2):213-8. doi: 10.1093/ageing/afu145. Epub 2014 Oct 16. PMID 25324330
- [Background] Jeffry S, Ruby C, Twersky J, Hanlon JT. Effect of an interdisciplinary team on suboptimal prescribing in a long-term care facility. The Consultant Pharmacist 14(12):1386-91, 1994.
- [Derived] Jungo KT, Deml MJ, Schalbetter F, Moor J, Feller M, Luthold RV, Huibers CJA, Sallevelt BTGM, Meulendijk MC, Spruit M, Schwenkglenks M, Rodondi N, Streit S. A mixed methods analysis of the medication review intervention centered around the use of the 'Systematic Tool to Reduce Inappropriate Prescribing' Assistant (STRIPA) in Swiss primary care practices. BMC Health Serv Res. 2024 Mar 18;24(1):350. doi: 10.1186/s12913-024-10773-y. PMID 38500163
- [Derived] Jungo KT, Weir KR, Cateau D, Streit S. Older adults' attitudes towards deprescribing and medication changes: a longitudinal sub-study of a cluster randomised controlled trial. BMJ Open. 2024 Jan 10;14(1):e075325. doi: 10.1136/bmjopen-2023-075325. PMID 38199626
- [Derived] Jungo KT, Ansorg AK, Floriani C, Rozsnyai Z, Schwab N, Meier R, Valeri F, Stalder O, Limacher A, Schneider C, Bagattini M, Trelle S, Spruit M, Schwenkglenks M, Rodondi N, Streit S. Optimising prescribing in older adults with multimorbidity and polypharmacy in primary care (OPTICA): cluster randomised clinical trial. BMJ. 2023 May 24;381:e074054. doi: 10.1136/bmj-2022-074054. PMID 37225248
- [Derived] Jungo KT, Meier R, Valeri F, Schwab N, Schneider C, Reeve E, Spruit M, Schwenkglenks M, Rodondi N, Streit S. Baseline characteristics and comparability of older multimorbid patients with polypharmacy and general practitioners participating in a randomized controlled primary care trial. BMC Fam Pract. 2021 Jun 22;22(1):123. doi: 10.1186/s12875-021-01488-8. PMID 34157981
- [Derived] Jungo KT, Rozsnyai Z, Mantelli S, Floriani C, Lowe AL, Lindemann F, Schwab N, Meier R, Elloumi L, Huibers CJA, Sallevelt BTGM, Meulendijk MC, Reeve E, Feller M, Schneider C, Bhend H, Burki PM, Trelle S, Spruit M, Schwenkglenks M, Rodondi N, Streit S. 'Optimising PharmacoTherapy In the multimorbid elderly in primary CAre' (OPTICA) to improve medication appropriateness: study protocol of a cluster randomised controlled trial. BMJ Open. 2019 Sep 3;9(9):e031080. doi: 10.1136/bmjopen-2019-031080. PMID 31481568
- See also: Project description by National Research Programme 74 "Smarter Healthcare" (NRP74) / Swiss National Science Foundation (SNSF) — http://www.nfp74.ch/de/projekte/ambulante-versorgung/projekt-rodondi